CLINICAL TRIAL: NCT03788525
Title: Reduction of Screen-Based Media Use in Families With Children: a Randomized Pilot Trial
Brief Title: Reduction of Screen-Based Media Use in Families With Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: European Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S-20170213; 716657 (Other Grant/Funding Number: European Research Council)
Record Dates: First submitted 2018-12-20; First posted 2018-12-27 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Feasibility Studies
Keywords: Screen time

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced recreational screen time (Experimental): Reducing recreational screen-based media use for a period of 2 weeks
  Interventions: Behavioral: Reduced recreational screen time
- Timed recreational screen time (Experimental): Reduced and timed recreational screen-based media use for a period of 2 weeks
  Interventions: Behavioral: Timed recreational screen time

INTERVENTIONS:
Behavioral: Reduced recreational screen time — Participants must remove all recreational screen-based media use beyond 3 hours/week. This includes all recreational screen-based media use inside and outside the household. As a tool to comply with the intervention the families will hand-over all portable screen-based media devices. In return, each participant who own a smartphone will receive a regular cell-phone which can only make phone calls and send text messages. For a maximum of ½ an hour a day, adult participants may use this device for necessary contact. The families are allowed a maximum of 3 hours/week of recreational screen time. If participants can not hand over their smartphones due to daily use for work purposes we will install an app tracking screen use on these devices.
  Arms: Reduced recreational screen time
Behavioral: Timed recreational screen time — Participants must remove all recreational screen-based media use after 6 PM. There are no restrictions on the amount of screen-based media use before 6 PM. Thus, before 6 PM, the participants must continue their habitual screen-based media use completely. However, after 6 PM, both work-related and recreational screen-based media use must be removed completely.
  Arms: Timed recreational screen time

SUMMARY:
The purpose of this pilot experiment is threefold.

1. To assess the efficacy of the recruitment strategy
2. To assess the acceptability and feasibility of the outcome measurement methods obtained in free-living in the participants homes
3. To assess the acceptability of the prescribed interventions to reduce screen media use

DETAILED DESCRIPTION:
Modern day's excessive use of screen-based media is heavily discussed in the public in terms of its possible harmful effects on physical and mental health among children and adults. To date there is little rigorously conducted research available on the effects of high use of todays screen-based media. Of particular notice, no controlled experimental studies in free-living have been carried out to study the immediate effects of screen-based media use on habitual physical activity patterns, sleep, and temporary stress- and emotional state.

To undertake a large-scale randomized controlled trial of the efficacy of limiting screen-based media use in families of parents and children the investigators aim to conduct a pilot study to assess the acceptability and feasibility of the outcome measurement methods obtained in free-living in the participants homes and the acceptability of the prescribed interventions to reduce screen media use. The investigators also perform the pilot study to investigate the efficacy of our recruitment strategy.

The participating families (households with children ≥4 and <18 years old) will be invited to answer a recruitment questionnaire sent out to their personal digital mailbox, which is a compulsory digital solution to receive mail from i.e. public authorities. Based on the survey answers eligible families (see section on inclusion/exclusion criteria) will be invited to participate in this pilot experiment. Families who are willing to participate will be randomized to one of two intervention groups after completion of the baseline measurement protocol. One group must reduce all recreational screen-based media use to less than three hours per week for a period of two weeks. Participants in this group will be asked to hand over their portable screen devices and in exchange they will be handed an old model Nokia phone. The other group must remove all screen-based media use (both work-related and recreational) after 6PM for a period of two weeks. The experiment does not include a control group. To ensure compliance to the interventions, the investigators will install an app, which will measure screen use on each participant's smartphone(s) and tablet(s). Furthermore, the investigators will connect a device to all televisions in each household, which will monitor television usage. To investigate the effect of the interventions all participants will go through a 7-day measurement protocol just before the family is randomized to one of the interventions and again during the last week of the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* High amount of screen-based media according to self-report (based on the adults only)
* In each household, at least one adult and one child must be above the 50th percentile for self-reported screen-based media use (characterized as "high" in this study). The 50th percentile is based on the responses from all adults who answered the recruitment survey.
* The children in the household are ≥ 4 and ≤ 18 years old, at the time the survey is sent out. In this way sleep measurements do not get distorted by infants and toddlers in the household (e.g. sleep).
* Adults and children who participate in the measurements must have the resources to remove all recreational- and work-/school-related screen-time in the evening hours, with a few exceptions, for a period of 2 weeks (intervention length).
* Participants must report that they consider the extent of their screen-based media use an issue
* Participants must report to be motivated to decrease screen-based media use for the whole family household.
* Family members who choose to not participate or are ineligible must be willing to support the success of this family experiment.

Exclusion Criteria:

* If the adults or children only reside in the household part time, i.e. have multiple addresses
* Diagnosis of stress from their general practitioner within the last year
* Diagnosis of sleep disorders from their general practitioner within the last year
* Working night shifts
* In any shape or form limited in one's ability to participate in habitual physical activity
* Has or is in inquiry of Neuropsychiatric disorders, such as Attention Deficit Hyperactivity Disorder (ADHD) or development disorders such as Autism.
* Already participating in research studies, such as the Odense Child Cohort

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Compliance to prescribed intervention (objective assessment) | 14 days (experiment period)
  Proportion of participants who are compliant to the prescribed intervention.
  Compliance is assessed objectively using data from the Device Tracker App (installed on all portable devices) and the television monitor installed on all televisions in the household.
Compliance to prescribed intervention (subjective assessment) | 14 days (experiment period)
  Proportion of participants who are compliant to the prescribed intervention.
  Compliance is assessed subjectively through a daily screen-media dairy. All participants are required to hold the daily screen-media dairy throughout the experiment period.

SECONDARY OUTCOMES:
Compliance to objective physical activity measurement | 14 days (experiment period)
  Proportion of participants wearing the accelerometer belts (Axivity AX3) for at least four out of seven measurements days at baseline and follow-up (at least one day must be a weekend day).
Compliance to sleep measurement | 14 days (experiment period)
  Proportion of participants wearing the sleep equipment (Zmachine Insight+) for at least two out of three measurement nights at baseline and follow-up.
Compliance to heart rate variability measurement | 14 days (experiment period)
  Proportion of participants wearing the heart rate variability device (Firstbeat Bodyguard 2) for at least two out of three measurement days at baseline and follow-up.
Compliance to saliva sampling protocol (only in adults) | 14 days (experiment period)
  Proportion of participants delivering salivary samples from two out of three measurement days which is equivalent to eight out of twelve samples at baseline and follow-up.
  Samples are collected by the participant at awakening, 30 min. after awakening, 45 min. after awakening, and just before bedtime.
Feasibility of the recruitment strategy | Up to four months
  Proportion of invited participants completing the full experiment period. Participants are invited and recruited continuously throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Grøntved, Ph.D., Principal Investigator — University of Southern Denamrk
Locations (1):
- University of Southern Denmark, Odense, Funen, Denmark

REFERENCES:
- [Result] Rasmussen MGB, Pedersen J, Olesen LG, Kristensen PL, Brond JC, Grontved A. Feasibility of two screen media reduction interventions: Results from the SCREENS pilot trial. PLoS One. 2021 Nov 15;16(11):e0259657. doi: 10.1371/journal.pone.0259657. eCollection 2021. PMID 34780511
- [Result] Sorensen SO, Pedersen J, Rasmussen MG, Kristensen PL, Grontved A. Feasibility of home-based sampling of salivary cortisol and cortisone in healthy adults. BMC Res Notes. 2021 Nov 2;14(1):406. doi: 10.1186/s13104-021-05820-4. PMID 34727972
- [Result] Pedersen J, Rasmussen M G B, Olesen L G, Kristensen P L, Grøntved A. Self-administered electroencephalography-based sleep assessment: compliance and perceived feasibility in children and adults. Sleep Science and Practice. 2021; 5(1):8. doi.org/10.1186/s41606-021-00059-1
- See also: Feasibility of two screen media reduction interventions: Results from the SCREENS pilot trial. PLoS One. 2021 Nov 15;16(11):e0259657. doi: 10.1371/journal.pone.0259657. eCollection — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0259657
- See also: Feasibility of home-based sampling of salivary cortisol and cortisone in healthy adults. BMC Res Notes. 2021 Nov 2;14(1):406. doi: 10.1186/s13104-021-05820-4. — https://bmcresnotes.biomedcentral.com/articles/10.1186/s13104-021-05820-4
- See also: Self-administered electroencephalography-based sleep assessment: compliance and perceived feasibility in children and adults. Sleep Science and Practice. 2021; 5(1):8. doi.org/10.1186/s4 — https://sleep.biomedcentral.com/articles/10.1186/s41606-021-00059-1